CLINICAL TRIAL: NCT06250946
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled, Parallel-group Phase ⅡStudy to Evaluate the Efficacy and Safety of HRS-7535 in Obese Subjects
Brief Title: Efficacy and Safety of HRS-7535 Tablets in Obese Subjects .
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HRS-7535-202
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A (Experimental): Subjects will receive escalated dose of HRS-7535 administered orally
  Interventions: Drug: HRS-7535;Placebo
- Group B (Experimental): Subjects will receive escalated dose of HRS-7535 administered orally
  Interventions: Drug: HRS-7535;Placebo
- Group C (Experimental): Subjects will receive escalated dose of HRS-7535 administered orally
  Interventions: Drug: HRS-7535;Placebo
- Group D (Experimental): Subjects will receive escalated dose of HRS-7535 administered orally
  Interventions: Drug: HRS-7535;Placebo
- Group E (Placebo Comparator): Subjects will receive Placebo administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS-7535;Placebo — HRS-7535;Placebo
  Arms: Group A; Group B; Group C; Group D
Drug: Placebo — Placebo
  Arms: Group E

SUMMARY:
The aim of this trial is to evaluate the efficacy and safety of HRS-7535 in Chinese Obese Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18-65 years of age at the time of signing informed consent;
2. At screening and random visit, 28.0 ≤BMI≤ 40.0 kg/m2;
3. Diet and exercise control for at least 3 months before screening and random visit, and less than 5 % self-reported change within the last 3 months.
4. Able and willing to provide a written informed consent

Exclusion Criteria:

1. Presence of clinically significant lab or ECG results that may affect the evaluation of the efficacy or safety of the study drug at screening visit;
2. Uncontrollable hypertension;
3. PHQ-9 score ≥15;
4. History of diabetes;
5. History of acute cardiovascular and cerebrovascular diseases within 6 months prior to screening;
6. Any organ-system malignancies developed within 5 years except for cured local basal cell cancer of the skin and in-situ cancer of the cervix;
7. Confirmed or suspected depression, bipolar disorder, suicidal tendencies, schizophrenia, or other serious mental illness;
8. Use of any medication or treatment that may have caused significant weight change within 2 months;
9. History of bariatric surgery;
10. history of blood donation or blood loss in the 3 months before screening, or blood transfusion in the 2 months before screening;
11. Surgery is planned during the trial;
12. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method;
13. Researchers and relevant staff of the research Centre or other people directly involved in the implementation of the programme, and their immediate family members.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight from baseline at Week 26 | Week 26

SECONDARY OUTCOMES:
Proportion of subjects with weight loss of ≥5%, ≥10%, ≥15% from baseline in body weight at Week 26 and Week 36 | Week 26 and Week 36
Percent change in body weight from baseline at Week 36 | Week 36
Change from baseline in body weight/ waist circumference/ BMI at Week 26 and Week 36 | Week 26 and Week 36
Change from baseline in Systolic blood pressure and diastolic blood pressure at Week 26 and Week 36 | Week 26 and Week 36
Change from baseline in fasting plasma glucoseat Week 26 and Week 36 | Week 26 and Week 36
Change from baseline in fasting serum insulin at Week 26 and Week 36 | Week 26 and Week 36
Change from baseline in HbA1c at Week 26 and Week 36 | Week 26 and Week 36
Change from baseline in total cholesterol (TC) at Week 26 and Week 36 | Week 26 and Week 36
Change from baseline in low density lipoprotein cholesterol (LDL-C) at Week 26 and Week 36 | Week 26 and Week 36
Change from baseline in high Density lipoprotein cholesterol (HDL-C) at Week 26 and Week 3 | Week 26 and Week 3
Change from baseline in triglycerides (TG) at Week 26 and Week 36 | Week 26 and Week 36

CONTACTS AND LOCATIONS:
Locations (1):
- The First Medical Center of Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided